CLINICAL TRIAL: NCT05168423
Title: Phase 1, Open-label Study Evaluating the Safety and Feasibility of CART-EGFR-IL13Ra2 Cells in Patients With EGFR-Amplified Recurrent Glioblastoma
Brief Title: CART-EGFR-IL13Ra2 in EGFR Amplified Recurrent GBM
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Kite Pharma (a Gilead Company) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16321
Record Dates: First submitted 2021-11-22; First posted 2021-12-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: 3+3 Dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Participants will receive a single fixed dose of 1x10^7 CART-EGFR-IL13Ra2 cells via intrathecal administration on Day 0.
  Interventions: Drug: CART-EGFR-IL13Ra2 Cells
- Cohort -1 (Experimental): Participants will receive a single fixed dose of 5x10^6 CART-EGFR-IL13Ra2 cells via intrathecal administration on Day 0.
  Interventions: Drug: CART-EGFR-IL13Ra2 Cells
- Cohort 2 (Experimental): Participants will receive a single fixed dose of 2.5x10^7 CART-EGFR-IL13Ra2 cells via intrathecal administration on Day 0.
  Interventions: Drug: CART-EGFR-IL13Ra2 Cells
- Cohort 3 (Experimental): Participants will receive a single fixed dose of 5x10^7 CART-EGFR-IL13Ra2 cells via intrathecal administration on Day 0.
  Interventions: Drug: CART-EGFR-IL13Ra2 Cells
- Cohort 4 (Experimental): Participants will receive two doses of CART-EGFR-IL13Rα2 cells, to determine the optimal dose schedule.
  Interventions: Drug: CART-EGFR-IL13Ra2 Cells

INTERVENTIONS:
Drug: CART-EGFR-IL13Ra2 Cells — autologous T cells transduced with a bicistronic lentiviral vector containing a murine scFv targeting EGFR and a humanized scFv targeting IL13Ra2

SUMMARY:
This is an open-label phase 1 study to assess the safety and feasibility of autologous T cells co-expressing two CARs targeting the cryptic EGFR epitope 806 and IL13Ra2 (referred to as "CART-EGFR-IL13Ra2 cells") in patients with EGFR-amplified glioblastoma, IDH-wildtype that has recurred following prior radiotherapy. This study will take place in two parts: an initial dose escalation phase followed by a dose exploration phase. In the dose expansion phase, the maximum tolerated dose (MTD) of CART-EGFR-IL13Ra2 cells will be determined using a standard 3+3 design. Once the MTD has been determined, the dose exploration phase will allow for further identification of a recommended dose for expansion (RDE) as well as the safety and feasibility of alternative dosing schedules.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written informed consent
2. Male or female age ≥ 18 years
3. Patients with glioblastoma, IDH-wildtype (as defined by WHO 2021 Classification of CNS Tumors) that has recurred following prior radiotherapy. For patients with tumors harboring methylation of the MGMT promoter, at least 12 weeks must have elapsed since completion of first-line radiotherapy.
4. Tumor tissue positive for wild-type EGFR amplification by NeoGenomics Laboratories. Archival tumor from patient's initial surgery at time of original diagnosis or recently collected tumor from time of recurrence are acceptable.
5. Surgical tumor resection for disease control/management or tumor biopsy to confirm tumor recurrence is clinically indicated in the opinion of the physician-investigator.
6. Adequate organ function defined as:

   1. Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 30 ml/min and not on dialysis.
   2. ALT/AST ≤ 3 x upper limit of normal range and total bilirubin ≤ 2.0 mg/dl, except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome (≤ 3.0 mg/dl).
   3. Left Ventricular Ejection Fraction (LVEF) ≥ 45% confirmed by ECHO/MUGA
   4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air
7. Karnofsky Performance Status ≥ 60%.
8. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Active hepatitis B or hepatitis C infection.
2. Any other active, uncontrolled infection.
3. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
4. Tumors primarily localized to the brain stem or spinal cord.
5. Severe, active co-morbidity in the opinion of the physician-investigator that would preclude participation in this study.
6. Receipt of bevacizumab within 3 months prior to physician-investigator confirmation of eligibility.
7. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10 mg daily of prednisone. Patients with autoimmune neurological diseases (such as MS or Parkinson's) will be excluded.
8. Patients who are pregnant or nursing (lactating).
9. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2039-12-19 (Estimated); Study Completion 2039-12-19 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with treatment related adverse events using NCI Common Terminology Criteria for Adverse Events (CTCAE) V5.0 | Up to 15 years following CART-EGFR-IL13Ra2 administration
  Type, frequency, severity, and attribution of adverse events
Number of subjects with dose-limiting toxicities (DLTs) | 28 days following initial treatment with CART-EGFR-IL13Ra2 cells
  Dose Escalation Phase only; Unacceptable toxicity as defined by the protocol
Determination of maximum tolerated dose (MTD). | 28 days following initial treatment with CART-EGFR-IL13Ra2 cellsnths
  Dose Escalation Phase only: The maximum tolerated dose (MTD) is defined as the highest dose explored at which 0 or 1 DLT occurs in 6 evaluable subjects.
Determine the recommended dose for expansion (RDE). | Up to 12 months following initial treatment with CART-EGFR-IL13Ra2 cells
Proportion of eligible subjects who receive all planned doses of CART-EGFR-IL13Ra2 cells. | 28 days following initial treatment with CART-EGFR-IL13Ra2 cells
  Cohort 4 only

SECONDARY OUTCOMES:
Proportion of subjects who enroll on this study who received study treatment. | 12 months
  Evaluated based on the proportion of subjects who screen fail and those who receive any dose of CART-EGFR-IL13Ra2 cells.
Frequency of manufacturing failures | 3 months
  Proportion of subjects with CART-EGFR-IL13Ra2 products that fail to meet the product release criteria, out of the number of subjects in whom manufacturing was attempted.
  Proportion of subjects with CART-EGFR-IL13Ra2 products that fail to meet the assigned dose, out of the number of subjects in whom manufacturing was attempted.
Progression-Free Survival (PFS) | Up to 15 years following CART-EGFR-IL13Ra2 administration
  Per modified RANO criteria
Objective Response Rate (ORR) | Up to 12 months following CART-EGFR-IL13Ra2 administration
  Per modified RANO criteria (in subjects with measurable disease at the time of study treatment); Proportion of subjects with confirmed CR and PR.
Duration of response (DOR) | Up to 15 years following initial CART-EGFR-IL13Ra2 administration
  Per modified RANO criteria (in subjects with measurable disease at the time of study treatment); Time from the date when a response of confirmed CR/PR is first met to the date of confirmed disease progression, death or receipt of alternative treatment other than CART-EGFR-IL13Ra2 retreatment.
Overall Survival (OS) | Up to 15 years following initial CART-EGFR-IL13Ra2 administration
  Time from initial study treatment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bagley, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bagley SJ, Desai AS, Fraietta JA, Silverbush D, Chafamo D, Freeburg NF, Gopikrishna GK, Rech AJ, Nabavizadeh A, Bagley LJ, Park J, Jarocha D, Martins R, Sarmiento N, Maloney E, Lledo L, Stein C, Marshall A, Leskowitz RM, Jadlowsky JK, Mackey S, Christensen S, Oner BS, Plesa G, Brennan A, Gonzalez V, Chen F, Barrett D, Colbourn R, Nasrallah MP, Mourelatos Z, Hwang WT, Alanio C, Siegel DL, June CH, Hexner EO, Binder ZA, O'Rourke DM. Intracerebroventricular bivalent CAR T cells targeting EGFR and IL-13Ralpha2 in recurrent glioblastoma: a phase 1 trial. Nat Med. 2025 Aug;31(8):2778-2787. doi: 10.1038/s41591-025-03745-0. Epub 2025 Jun 1. PMID 40451950
- [Derived] Bagley SJ, Logun M, Fraietta JA, Wang X, Desai AS, Bagley LJ, Nabavizadeh A, Jarocha D, Martins R, Maloney E, Lledo L, Stein C, Marshall A, Leskowitz R, Jadlowsky JK, Christensen S, Oner BS, Plesa G, Brennan A, Gonzalez V, Chen F, Sun Y, Gladney W, Barrett D, Nasrallah MP, Hwang WT, Ming GL, Song H, Siegel DL, June CH, Hexner EO, Binder ZA, O'Rourke DM. Intrathecal bivalent CAR T cells targeting EGFR and IL13Ralpha2 in recurrent glioblastoma: phase 1 trial interim results. Nat Med. 2024 May;30(5):1320-1329. doi: 10.1038/s41591-024-02893-z. Epub 2024 Mar 13. PMID 38480922